CLINICAL TRIAL: NCT03155217
Title: Safety of Targeted Therapies in Elderly Patients (Over 5 and 75 Year-old) With Metastatic Melanoma
Brief Title: Tolerance of Targeted Therapy Used in Metastatic Melanoma in Patients Aged Over 65 and 75-year-old
Acronym: TOLBRIPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0048
Record Dates: First submitted 2017-05-05; First posted 2017-05-16 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; elderly; tolerance; adverse effects; targeted therapies
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients over 75 years: Patients with MM treated with single or combination therapy over 75 years of age.
- patients between 65 and 75 years: Patients aged 65-75 years with MM treated with single or dual therapy
- patients less than 65 years: patients less than 65 years with MM treated with single or dual therapy

SUMMARY:
Since 2013, therapeutic care of metastatic melanoma (MM) has greatly improved, especially thanks to BRAF and MEK targeted therapies. The efficacy of these treatments that are now used daily at first line for BRAF mutated MM is widely approved. Their toxicities, in monotherapy or in association, are also well-known: fever, arthralgias, digestive disorders, cutaneous rash, fatigue, photosensitivity, alopecia, cutaneous hyperkeratosis, squamous cell carcinomas, keratoacanthomas, de novo melanomas… However, onco-dermatologists are more and more faced with MM of elderly patients. Indeed, life expectancy continues to increase and the over-75-year-old age group is becoming larger. These patients are still active but much more vulnerable. Nevertheless, there is no data in the literature for this fragile population except the MM pivotal studies subgroups of those over 65-year-old. The results vary with different regimens. Therefore, there is a wide lack of information that could help make a therapeutic decision, inform patients, prevent or treat side effects of BRAF and MEK inhibitors in elderly patients

DETAILED DESCRIPTION:
Since 2013, therapeutic care of metastatic melanoma (MM) has greatly improved, especially thanks to BRAF and MEK targeted therapies. The efficacy of these treatments that are now used daily at first line for BRAF mutated MM is widely approved. Their toxicities, in monotherapy or in association, are also well-known: fever, arthralgias, digestive disorders, cutaneous rash, fatigue, photosensitivity, alopecia, cutaneous hyperkeratosis, squamous cell carcinomas, keratoacanthomas, de novo melanomas… However, onco-dermatologists are more and more faced with MM of elderly patients. Indeed, life expectancy continues to increase and the over-75-year-old age group is becoming larger. These patients are still active but much more vulnerable. Nevertheless, there is no data in the literature for this fragile population except the MM pivotal studies subgroups of those over 65-year-old. The results vary with different regimens. Therefore, there is a wide lack of information that could help make a therapeutic decision, inform patients, prevent or treat side effects of BRAF and MEK inhibitors in elderly patients. This work aims to study the targeted therapies tolerance in over 65 or 75-year-old patients with BRAF mutated MM. The French clinical and biological database MELBASE will be analysed to carry out a descriptive retrospective multicentric study. This real-life assessment of the adverse effects in older patients will result in more adapted therapeutic decisions, better informed patients and improved follow-up care in order to increase quality of life and life expectancy.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic melanoma

Exclusion Criteria:

* none

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: More 65 and 75 yo patients, Braf mutated, treated with targeted therapies in mono or bitherapy for metastatic melanoma
Sampling Method: Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
grade 3-4 adverse effects | 1 day
  Analyze the relationship between Grade 3 and Level 4 adverse events in subjects older than 65 or 75 years of age compared to patients under 65 years of age

SECONDARY OUTCOMES:
Treatment modification | 1 day
  Analyze treatment changes with progression-free survival and overall follow-up in patients over 65 or 75 years of age compared to patients younger than 65 years.

CONTACTS AND LOCATIONS:
Overall Officials: ondine BECQUART, Study Chair — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided